CLINICAL TRIAL: NCT03790488
Title: Phase 1 First in Human Study of Programmed Cell Death Receptor-1 (PD-1) Inhibitor Monoclonal Antibody (mAb) JTX-4014 in Adult Subjects With Advanced Refractory Solid Tumor Malignancies
Brief Title: Study of a PD-1 Inhibitor (JTX-4014) in Subjects With Solid Tumor Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jounce Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JTX-4014-101
Record Dates: First submitted 2018-12-21; First posted 2018-12-31 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Cancer
Keywords: Solid Tumor Malignancies; JTX-4014; Monoclonal Antibody (mAb); Programmed Cell Death Receptor-1 (PD-1); Immunotherapy; Immuno-oncology; Dose Escalation
MeSH Terms: conditions — Neoplasms | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JTX-4014 (Experimental): Phase 1 dose escalation of PD-1 inhibitor mAb JTX-4014 by intravenous infusion
  Interventions: Drug: JTX-4014

INTERVENTIONS:
Drug: JTX-4014 — Specified dose on specified days
  Other Names: PD-1 Inhibitor

SUMMARY:
JTX-4014-101 is a Phase 1, open label, dose escalation clinical study of JTX-4014 in adult subjects with advanced refractory solid tumor malignancies, to determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D).

DETAILED DESCRIPTION:
JTX-4014 is a fully human IgG4 monoclonal antibody designed to specifically bind to PD-1 and block its interaction with its ligands, PD-L1 and PD-L2, to augment anti-tumor T cell activity. This is a Phase 1, first in human, open label, multicenter, dose escalation clinical study to evaluate the safety, tolerability, and PK of JTX-4014 when administered as a single agent to adult subjects with advanced refractory solid tumor malignancies. The intent of this study will be to determine the MTD and RP2D.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to participate and comply with all study requirements and provide signed and dated informed consent prior to initiation of any study procedures;
2. Histologically or cytologically confirmed extracranial solid tumor malignancy that is recurrent, metastatic, or persistent after at least 1 line of standard therapy and with no further standard treatment options that are likely to provide meaningful clinical benefit;
3. Evaluable or measurable disease, according to the RECIST version 1.1, that has objectively progressed since (or on) previous treatment as assessed by the Investigator; while target lesions are not required, target lesions should be measured if present;
4. ≥ 18 years of age;
5. ECOG performance status 0 or 1;
6. Predicted life expectancy of ≥ 3 months;
7. Have laboratory values (obtained ≤ 28 days prior to first infusion day) in accordance with the study protocol;
8. For women of childbearing potential (WOCBP): negative serum pregnancy test within 72 hours prior to planned Cycle 1 Day 1 (C1D1) and a negative urine pregnancy test on C1D1;
9. WOCBP and males whose partners are WOCBP must agree to use a highly effective method of birth control throughout their participation and for 5 months following the last study drug administration;
10. Subjects with medical history of the following must be discussed with the Medical Monitor:

    1. Prior biliary tract disorders (as based on hepatobiliary system organ class high level terms of: obstructive bile duct disorders, hepatic vascular disorders, structural and other bile duct disorders).
    2. Portal hypertension and/or hepatic vascular disorders.

Exclusion Criteria:

1. Concurrent anticancer treatment, either FDA-approved, palliative, or investigational for the cancer being evaluated in this study or for other cancers (with protocol-specified exceptions);
2. Prior receipt of a PD-1 or PD-L1 inhibitor mAb, including JTX-4014;
3. The therapies listed below within the specified timeframe or ongoing toxicity attributed to prior therapy that was > Grade 1 according to the NCI CTCAE, with protocol-specified exceptions:

   1. Major surgery < 4 weeks prior to planned C1D1;
   2. Biologic therapy, including non-PD-1/PD-L1 inhibitor immunotherapy, < 28 days prior to planned C1D1;
   3. Chemotherapy < 21 days prior to planned C1D1, or < 42 days for mitomycin or nitrosoureas;
   4. Targeted small molecule therapy < 14 days prior to planned C1D1;
   5. Hormonal or other adjunctive therapy for cancers other than the cancer under evaluation in this study that started < 14 days prior to planned C1D1, with protocol-specified exceptions;
   6. Radiation therapy < 21 days prior to planned C1D1, with protocol-specified exceptions;
   7. Any prior organ transplantation, including allogeneic or autologous stem cell transplantation;
4. History of intolerance, hypersensitivity, or treatment discontinuation due to severe immune-related adverse events on prior non PD 1/PD L1 inhibitor immunotherapy;
5. Diagnosis of immunodeficiency, either primary or acquired, or treatment with immunosuppressive levels of systemic corticosteroids or any other form of immunosuppressive therapy within 7 days prior to planned C1D1, with protocol-specified exceptions;
6. Known severe intolerance or life-threatening hypersensitivity reactions to humanized mAbs or intravenous immunoglobulin preparations; any history of anaphylaxis; prior history of human anti-human antibody response; known allergy to any of the study medications, their analogues, or excipients;
7. Symptomatic or uncontrolled brain metastases, leptomeningeal disease, or spinal cord compression not definitively treated with surgery or radiation, with protocol-specified exceptions;
8. Active and clinically relevant bacterial, fungal, or viral infection, including known hepatitis A, B, C, or human immunodeficiency virus;
9. Receipt of live vaccines within 30 days of planned C1D1;
10. Women who are pregnant or breastfeeding or who plan to become pregnant/breastfeed while on study; men who plan to father children during the study;
11. History of pneumonitis requiring treatment with corticosteroids, interstitial lung disease, or severe radiation pneumonitis (excluding localized radiation pneumonitis);
12. Symptomatic ascites or pleural effusion;
13. History of acute diverticulitis, intra-abdominal abscess, gastrointestinal obstruction, or abdominal carcinomatosis;
14. Symptomatic cardiac or cerebrovascular disease that is unresponsive to surgical or medical management;
15. Medical or social condition that, in the opinion of the Investigator, might place the subject at increased risk, adversely affect compliance, or confound safety or other clinical study data interpretation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
% subjects with adverse events (AEs) | Approximately 12 months
% subjects with serious adverse events (SAEs) | Approximately 12 months
% subjects with dose-limiting toxicities (DLTs) | Approximately 12 months
% subjects with changes from baseline in pro-inflammatory cytokines | Approximately 12 months
% subjects with clinically significant change from baseline in clinical laboratory tests | Approximately 12 months
Maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of JTX-4014 | Approximately 12 months

SECONDARY OUTCOMES:
Maximum measured concentration in serum (Cmax) | Approximately 12 months
Time from dosing to Cmax (Tmax) | Approximately 12 months
Area under the serum concentration-time curve (AUC) | Approximately 12 months
Last measurable concentration (Clast) | Approximately 12 months
Time to last measurable concentration (Tlast) | Approximately 12 months
Terminal half-life (t1/2) | Approximately 12 months
Accumulation ratio of JTX-4014 | Approximately 12 months
Evaluate anti-drug antibodies (ADA) against JTX-4014 | Approximately 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stew Kroll, Study Director — Jounce Therapeutics, Inc.
Locations (4):
- United States (4):
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Florida Cancer Specialists - Sarasota Cattlemen, Sarasota, Florida
  - START Midwest - Cancer & Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Papadopoulos KP, Lakhani N, Falchook GS, Riley G, Baeck J, Brown KS, Gordon G, Le L, Wang JS. Phase I, first-in-human trial of programmed cell death receptor-1 (PD-1) inhibitor, JTX-4014, in adult patients with advanced, refractory, solid tumors. Cancer Immunol Immunother. 2021 Mar;70(3):763-772. doi: 10.1007/s00262-020-02730-5. Epub 2020 Sep 28. PMID 32989552